CLINICAL TRIAL: NCT02636322
Title: A Phase II Study of Rituximab, Lenalidomide, and Ibrutinib Combined With Chemotherapy for Patients With High Risk Diffuse Large B-Cell Lymphoma
Brief Title: Smart Start: A Phase II Study of Rituximab, Lenalidomide, and Ibrutinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0147; NCI-2016-00017 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0147 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Diffuse Large B-Cell Lymphoma Unclassifiable
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin; Etoposide; ibrutinib; Lenalidomide; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RLI WITH EPOCH (Experimental): SMART START: Patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  After SMART START therapy, patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Patients also receive etoposide IV over 24 hours on days 1-4, prednisone PO QD on days 1-5, vincristine sulfate IV over 24 hours on days 1-4, doxorubicin hydrochloride IV over 24 hours on days 1-4, and cyclophosphamide IV over 1 hour on day 5. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Ibrutinib; Drug: Lenalidomide; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate
- RLI WITH R-CHOP (Experimental): SMART START: Patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  After SMART START therapy, patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Patients also receive prednisone PO QD on days 1-5, vincristine sulfate IV over 1 hour on day 1, doxorubicin hydrochloride IV over 1 hour on day 1, and cyclophosphamide IV over 1 hour on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin Hydrochloride; Drug: Ibrutinib; Drug: Lenalidomide; Drug: Prednisone; Biological: Rituximab; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
  Arms: RLI WITH EPOCH
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II trial studies how well giving rituximab, lenalidomide, and ibrutinib with chemotherapy works in treating patients with high-risk diffuse large B-cell lymphoma. High-risk large B-cell lymphoma is a type of cancer of the immune system that is usually fast-growing in the body. Monoclonal antibodies, such as rituximab, may block cancer growth in different ways by targeting certain cells. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as lenalidomide, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as etoposide, prednisone, vincristine sulfate, cyclophosphamide, and doxorubicin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving rituximab, ibrutinib, and lenalidomide with combination chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rate at the end of 2 cycles of therapy with rituximab, lenalidomide, and ibrutinib in patients with high risk newly diagnosed non-germinal center B-cell-like diffuse large B-cell lymphoma (non-GCB DLBCL).

II. To determine the complete response rate at the end of 6 cycles of therapy with rituximab, lenalidomide, and ibrutinib combined with chemotherapy (cyclophosphamide, doxorubicin hydrochloride [hydroxydaunorubicin hydrochloride], vincristine sulfate [Oncovin], prednisone [CHOP] or etoposide, prednisone, vincristine sulfate [Oncovin], cyclophosphamide, doxorubicin hydrochloride [hydroxydaunorubicin hydrochloride] [EPOCH]) in patients with high risk newly diagnosed non-GCB DLBCL.

SECONDARY OBJECTIVES:

I. To determine the overall response rate, landmark survival outcomes (progression free and overall survival), and safety of lenalidomide and ibrutinib with chemotherapy (CHOP or EPOCH) in patients with high risk newly diagnosed non-GCB DLBCL.

II. To evaluate descriptively the complete response rate in rituximab, lenalidomide, ibrutinib (RLI)-CHOP and in RLI-EPOCH.

EXPLORATORY OBJECTIVES:

I. To evaluate the baseline and therapy induced changes in the profile of mutations, gene expression, minimal residual disease clonotype levels, immune cell subsets, and tumor protein expression in tumor biopsy and blood samples in patients with high risk newly diagnosed non-GCB DLBCL.

OUTLINE:

SMART START: Patients receive rituximab intravenously (IV) over 4-6 hours on day 1, lenalidomide orally (PO) once daily (QD) on days 1-10, and ibrutinib PO QD on days 1-21. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity.

RLI WITH EPOCH: After SMART START therapy, patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Patients also receive etoposide IV over 24 hours on days 1-4, prednisone PO QD on days 1-5, vincristine sulfate IV over 24 hours on days 1-4, doxorubicin hydrochloride IV over 24 hours on days 1-4, and cyclophosphamide IV over 1 hour on day 5. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

RLI WITH R-CHOP: After SMART START therapy, patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Patients also receive prednisone PO QD on days 1-5, vincristine sulfate IV over 1 hour on day 1, doxorubicin hydrochloride IV over 1 hour on day 1, and cyclophosphamide IV over 1 hour on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, and then every 4 months for another year.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of previously untreated DLBCL of the non-GCB DLBCL subtype
* No prior treatment except a prior limited-field radiotherapy, a short course of glucocorticoids =< 25 mg daily of prednisone equivalent which must cease prior to day 1 of cycle 1, and/or cyclophosphamide for an urgent lymphoma related problem at diagnosis (e.g. epidural cord compression, superior vena cava syndrome)
* Patient or durable power of attorney (DPA) for healthcare must be able to understand and voluntarily sign an Institutional Review Board (IRB) -approved informed consent form
* Patients must have bi-dimensional measurable disease, as defined as radiographically apparent disease with the longest dimension of >= 1.5 cm
* Patients with performance status of =< 3 (3 only allowed if decline in status is deemed related to lymphoma and felt potentially reversible by the treating physician)
* Serum bilirubin < 1.5 x upper limit of normal (ULN) except in patients with Gilbert's syndrome as defined by > 80% unconjugated bilirubin
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN or < 5 x ULN if hepatic metastases are present
* Absolute neutrophil count (ANC) > 1000/mm^3 unless deemed related to lymphoma involvement in the bone marrow and felt potentially reversible by the treating physician
* Platelets > 100,000/mm^3 unless deemed related to lymphoma involvement in the bone marrow and felt potentially reversible by the treating physician
* Renal function assessed by calculated creatinine clearance:

  * Calculated creatinine clearance >=30 ml/min by Cockcroft-Gault formula
* Patients must be willing to receive transfusions of blood products
* All study participants must be registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS) program, and be willing and able to comply with the requirements of the REMS program
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening and must adhere to the scheduled pregnancy testing as required in the Revlimid REMS program
* Women of childbearing potential and men who are sexually active with a woman of childbearing potential must be practicing a highly effective method of birth control during and after the study (12 months for women and 3 months for men), consistent with local regulations regarding the use of birth control methods for subjects participating in this clinical study; men must agree to not donate sperm during and for up to 3 months after their conclusion of therapy on study
* Able to take aspirin (81 mg) daily or alternative therapy as prophylactic anticoagulation

Exclusion Criteria:

* Any serious medical condition including but not limited to uncontrolled hypertension, uncontrolled congestive heart failure within past 6 months prior to screening (class 3 [moderate] or class 4 [severe] cardiac disease as defined by the New York Heart Association Functional Classification), uncontrolled diabetes mellitus, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), left ventricular ejection fraction (LVEF) less than 40%, renal failure, active infection, history of invasive fungal infection, moderate to severe hepatic disease (Child Pugh class B or C), active hemorrhage, laboratory abnormality, or psychiatric illness that, in the investigators opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form; patients with history of cardiac arrhythmias should have cardiac evaluation and clearance
* Pregnant or lactating females
* Known hypersensitivity to lenalidomide or thalidomide, ibrutinib, rituximab, etoposide, vincristine, doxorubicin, cyclophosphamide, or prednisone
* Known human immunodeficiency virus (HIV) infection; patients with active hepatitis B infection (not including patients with prior hepatitis B vaccination; or positive serum hepatitis B antibody); known hepatitis C infection is allowed as long as there is no active disease and is cleared by gastrointestinal (GI) consultation
* All patients with central nervous system involvement with lymphoma
* Diagnosis of prior malignancy within the past 2 years with the exception of successfully treated basal cell carcinoma, squamous cell carcinoma of the skin, carcinoma "in situ" of the cervix or breast; history of other malignancies are allowed if in remission (including prostate cancer patients in remission from radiation therapy, surgery or brachytherapy), not actively being treated, with a life expectancy > 3 years
* Significant neuropathy (grades 2 or grade 1 with pain) within 14 days prior to enrollment
* Contraindication to any of the required concomitant drugs or supportive treatments or intolerance to hydration due to preexisting pulmonary or cardiac impairment including pleural effusion requiring thoracentesis or ascites requiring paracentesis not due to lymphoma
* Patients with active pulmonary embolism or deep vein thrombosis (diagnosed within 30 days of study enrollment)
* Patients with severe bradycardia (heart rate < 40 beats per minute [bpm], hypotension, light-headedness, syncope)
* Major surgery within 4 weeks of study entry, or wound that is not healed from prior surgery or trauma
* History of stroke or intracranial hemorrhage within 6 months prior to study entry
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires chronic treatment with strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors
* Vaccinated with live, attenuated vaccines within 4 weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Westin J, Davis RE, Feng L, Hagemeister F, Steiner R, Lee HJ, Fayad L, Nastoupil L, Ahmed S, Rodriguez A, Fanale M, Samaniego F, Iyer SP, Nair R, Oki Y, Fowler N, Wang M, Ma MCJ, Vega F, McDonnell T, Pinnix C, Griffith D, Lu Y, Tewari S, Sun R, Scott DW, Flowers CR, Neelapu S, Green MR. Smart Start: Rituximab, Lenalidomide, and Ibrutinib in Patients With Newly Diagnosed Large B-Cell Lymphoma. J Clin Oncol. 2023 Feb 1;41(4):745-755. doi: 10.1200/JCO.22.00597. Epub 2022 Aug 11. PMID 35952327
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: for testing in up to 60 patients with newly diagnosed ABC DLBCL. Patients will start with RLI alone prior to the use of chemotherapy ("Smart Start") for ≤2 cycles, followed by 6 cycles of RLI with dose adjusted (DA) EPOCH.
Groups:
- RLI WITH EPOCH/RCHOP: SMART START: Patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  After SMART START therapy, patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Patients also receive prednisone PO QD on days 1-5, vincristine sulfate IV over 1 hour on day 1, doxorubicin hydrochloride IV over 1 hour on day 1, and cyclophosphamide IV over 1 hour on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | RLI WITH EPOCH/RCHOP
Started | 58
Complete Response | 21
Partial Response | 29
Non Responsive | 8
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- RLI WITH EPOCH/R-CHOP: SMART START: Patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  After SMART START therapy, patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Patients also receive etoposide IV over 24 hours on days 1-4, prednisone PO QD on days 1-5, vincristine sulfate IV over 24 hours on days 1-4, doxorubicin hydrochloride IV over 24 hours on days 1-4, and cyclophosphamide IV over 1 hour on day 5. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  Patients also receive prednisone PO QD on days 1-5, vincristine sulfate IV over 1 hour on day 1, doxorubicin hydrochloride IV over 1 hour on day 1, and cyclophosphamide IV over 1 hour on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
Arm/Group | RLI WITH EPOCH/R-CHOP
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 28
Age, Continuous [Median (Full Range); unit: Years] | 63.5 [29 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 47
  More than one race | 7
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: After two cycles of RLI
Time Frame: Up to 42 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RLI With EPOCH/CHOP: SMART START: Patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity.
  After SMART START therapy, patients receive rituximab IV over 4-6 hours on day 1, lenalidomide PO QD on days 1-10, and ibrutinib PO QD on days 1-21. Patients also receive prednisone PO QD on days 1-5, vincristine sulfate IV over 1 hour on day 1, doxorubicin hydrochloride IV over 1 hour on day 1, and cyclophosphamide IV over 1 hour on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
Arm/Group | RLI With EPOCH/CHOP
Number analyzed (Participants) | 58
percentage of participants | 86.2 [74.6 to 93.9]

2. Primary Outcome: Overall Response Rate
Description: After two cycles of RLI plus two cycles of RLI-chemotherapy
Time Frame: up to 84 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RLI With EPOCH/CHOP
Number analyzed (Participants) | 58
percentage of participants | 100 [93.6 to 100]

3. Secondary Outcome: Progression Free Survival at 2 Years
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RLI With EPOCH/CHOP
Number analyzed (Participants) | 58
percentage of participants | 91.3 [84.3 to 98.9]

4. Secondary Outcome: Overall Survival for 2 Years
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | RLI WITH EPOCH/RCHOP
Number analyzed (Participants) | 58
Participants | 58

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | RLI WITH EPOCH/R-CHOP
All-Cause Mortality (participants affected / at risk) | 2/60
Serious Adverse Events (participants affected / at risk) | 24/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RLI WITH EPOCH/R-CHOP (N=60)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Acute Kidney injury (Renal and urinary disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial fibrilation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood and Lymphatic other lymphoma tumor abscess, axilla (Blood and lymphatic system disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 24 (31)
Fever (General disorders) | 7 (8)
Infections and infestations - Other, Acute kidney infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, Bacteremia (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (3)
Memory impairment (Nervous system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Multi-organ failure (General disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (5)
Non-cardiac chest pain (General disorders) | 1 (1)
Platelet count decrease (Investigations) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin and subcutaneous Cellulitis right foot (Skin and subcutaneous tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 5 (5)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
White blood cell decrease (Investigations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RLI WITH EPOCH/R-CHOP (N=60)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Acute Kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (15)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Amnesia (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 42 (141)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 8 (8)
Artrial fibliration (Cardiac disorders) | 5 (6)
Atrial Flutter (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (8)
Bacteremia (Infections and infestations) | 1 (1)
Bladder infection (Renal and urinary disorders) | 1 (2)
Blood bilirubin increase (Investigations) | 4 (5)
Blurred vision (Eye disorders) | 21 (23)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Cardiac disorders - Other, specify increase heart rate (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 42 (54)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Creatinine increase (Investigations) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 47 (81)
Dizziness (Nervous system disorders) | 32 (38)
Dry Eye (Eye disorders) | 17 (18)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26 (32)
Dysuria (Renal and urinary disorders) | 1 (1)
"Ear and labyrinth disorders - Other Ear discharge bilateral" (Ear and labyrinth disorders) | 1 (1)
Edema face (General disorders) | 2 (2)
Edema Limbs (General disorders) | 30 (38)
Edema trunk (General disorders) | 1 (2)
Endocrine disorder Polydipsia (Endocrine disorders) | 1 (1)
Endocrine disorder Polyuria (Endocrine disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Eye disorder Blepharitis of right eye (Eye disorders) | 1 (1)
Eye disorder light sensitivity (Eye disorders) | 1 (1)
Eye infection (Eye disorders) | 1 (1)
Facila pain (General disorders) | 1 (1)
Fatigue (General disorders) | 58 (80)
Febrile Neutorpenia (Blood and lymphatic system disorders) | 2 (2)
Fever (General disorders) | 20 (23)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Gastrointestinal disorders - Other, Ulcer on left oral cavity (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, bloody stool (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, indigestion (Gastrointestinal disorders) | 1 (1)
Generalized edema (General disorders) | 1 (1)
Headache (Nervous system disorders) | 13 (17)
Hematuria (Renal and urinary disorders) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hoarseness (Reproductive system and breast disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypercalcemia (Investigations) | 2 (2)
Hyperglycemia (Investigations) | 1 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperuricemia (Investigations) | 1 (1)
Hypoalbuminemia (Investigations) | 2 (2)
Hypocalcemia (Investigations) | 2 (5)
Hypokalemia (Investigations) | 13 (31)
Hypomagnesemia (Investigations) | 7 (8)
Hyponatremia (Investigations) | 7 (10)
Hypophosphatemia (Investigations) | 6 (12)
Hypotension (Vascular disorders) | 4 (4)
Ileus (Vascular disorders) | 1 (1)
Infections and infestations others right great toe (Infections and infestations) | 2 (2)
Infections and infestations others (Infections and infestations) | 1 (1)
Infections other Clostridium Difficile infection (Infections and infestations) | 1 (1)
Infections and infestations others vaginal yeast (Infections and infestations) | 1 (1)
Infections and infestations others Coronavirus (Infections and infestations) | 1 (1)
Infections and infestations others Oral Candidiasis (Infections and infestations) | 1 (1)
Infections and infestations others left great toe (Infections and infestations) | 1 (1)
insomnia (Psychiatric disorders) | 9 (9)
Leukocytosis (Blood and lymphatic system disorders) | 2 (5)
Localized edema (General disorders) | 1 (1)
lung infection (Reproductive system and breast disorders) | 1 (1)
memory impairment (Psychiatric disorders) | 23 (23)
Metabolism and nutrition disorders other diaphoresis (Metabolism and nutrition disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 45 (61)
Musculoskeletal and connective tissue disorder - Other, Restless leg syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other,Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Hand cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 35 (45)
Nasal congestionres (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 51 (72)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms Benign, Malignant and Unspecified (Incl Cysts and Polyps) Left thigh nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nervous system disorders - Other, neck stiffness (Nervous system disorders) | 1 (1)
Neutrophil count decrease (Investigations) | 36 (95)
Non-cardiac chest pain (General disorders) | 2 (2)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Pain extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 4 (4)
Palpatations (Cardiac disorders) | 3 (4)
Paronychia (Infections and infestations) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 49 (78)
Pharyngitis (Gastrointestinal disorders) | 1 (1)
Platelet count decrease (Investigations) | 40 (146)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 (5)
presyncope (Nervous system disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 11 (15)
rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 (26)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal Pain (Gastrointestinal disorders) | 1 (1)
Reproductive System and Breast Disorders vaginal bleeding (Reproductive system and breast disorders) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracicand mediastinal disorder thoat pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracicand mediastinal disorder Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis infective (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Sepsis (Infections and infestations) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Skin and subcutaneous tissue disorders Fungal rash on feet (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders left areola redness (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders blisters on hands and feet bilateral (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders itchy scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders rash on torso and feet (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders Scalp tenderness (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Gastrointestinal disorders) | 3 (3)
Superior vena cava syndrome (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 5 (5)
upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 8 (11)
Vaginal infection (Reproductive system and breast disorders) | 1 (1)
Vascular access complication (Vascular disorders) | 1 (1)
vascular other Thrombus non occlusive (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 21 (24)
Watering eyes (Eye disorders) | 14 (14)
Weight loss (Investigations) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT02636322/Prot_SAP_000.pdf